CLINICAL TRIAL: NCT02295566
Title: RATNO (Reducing Antibiotic Tolerance Using NO) Reducing Antibiotic Tolerance Using Low Dose Nitric Oxide in Cystic Fibrosis - a Phase 2 Pilot Study
Brief Title: RATNO, Reducing Antibiotic Tolerance Using Nitric Oxide in CF - a Phase 2 Pilot Study
Acronym: RATNO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Collaborators: University of Southampton (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RHM CHI0548; 2010-023529-39 (EudraCT Number); 11/H0502/7 (Other: National Research Ethics Service)
Record Dates: First submitted 2014-08-20; First posted 2014-11-20 (Estimated); Last update posted 2024-05-30 (Actual); Status verified 2014-11

CONDITIONS: Cystic Fibrosis
Keywords: Nitric Oxide; Pseudomonas Aeruginosa; Biofilm
MeSH Terms: conditions — Cystic Fibrosis; Pseudomonas Infections | interventions — Nitric Oxide; Air; Oxygen

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nitric Oxide Group (Active Comparator): Inhaled Nitric Oxide delivered via nasal canulae at 10ppm for 8 hours a night for 7 nights.
  Interventions: Drug: Nitric Oxide
- Control Group (Placebo Comparator): Air/oxygen mix (according to clinical need) delivered via nasal canulae for 8 hours a night for 7 nights.
  Interventions: Drug: Control

INTERVENTIONS:
Drug: Nitric Oxide — Not required
  Arms: Nitric Oxide Group
Drug: Control — Not required
  Other Names: Air; Oxygen
  Arms: Control Group

SUMMARY:
The lungs of most patients with cystic fibrosis (CF) become chronically infected with bacteria called Pseudomonas aeruginosa during childhood. This infection is now known to consist of free-living bacteria (known as "planktonic bacteria") and bacteria in colonies on body surfaces known as "biofilms". The bacteria in biofilms are more resistant and tolerant to antibiotics. Current CF treatment of exacerbations aims to eradicate or control pseudomonal infection using aggressive antibiotic regimes.

Despite this treatment many patients develop chronic infection which is never cleared. Chronic infection causes damage to the lungs. Patients colonised with Pseudomonas are more unwell and die at a younger age. Our laboratory has established that low dose nitric oxide (NO) can disrupt pseudomonal biofilms in the laboratory. This pilot study will discover whether non-toxic levels of NO administered to participants during an episode of acute infection (exacerbation) will disrupt bacteria from biofilms and increase the effectiveness of antibiotic therapy. This protocol describes a participant-blind randomised controlled pilot study of treatment with nitric oxide gas during an acute infective exacerbation (also known simply as an "acute exacerbation"). Patients with CF aged 12 or above will be asked to take part.

They will be randomised to receive 7 days either of inhaled nitric oxide gas or placebo alongside standard therapy during an exacerbation. Sputum samples will be obtained before, during and after the treatment period for microbiological analysis. The primary endpoint will be the microbiological effect on bacterial biofilms before and after NO adjunctive therapy. Secondary microbiological endpoints will include the between group differences in pseudomonal colony forming units (CFU"s), biofilm NO levels and detailed characterisation of biofilms before and after treatment.

Secondary clinical endpoints will include lung function and well-established indicators quality of life. The aim of this randomised pilot study is as proof of concept and to guide the design of a large multi-centre trial to definitively evaluate the effectiveness of NO or NO donors as adjunctive therapy in CF.

DETAILED DESCRIPTION:
Not required

ELIGIBILITY:
Inclusion Criteria:

* Adolescents and young adults with cystic fibrosis aged 12 or above
* Colonised with Pseudomonas aeruginosa (confirmed on sputum sample)

Exclusion Criteria:

* Colonisation with Burkholderia cepacia
* Known hypersensitivity to the antibiotics used in the study
* Other known contraindications to the antibiotics to be used in the study including known aminoglycoside related hearing/renal damage
* Patients requiring non-invasive ventilation (NIV)
* Patients who have a pneumothorax
* Patients who are admitted for specific treatment of nontuberculous mycobacteria (NTM)
* Patients who cannot tolerate nasal cannula e.g. those who cannot breathe through their nose
* Patients who have nasal polyposis that is causing significant blockage of the nasal passages
* Adolescents who are not Gillick competent (and therefore not able to give their own assent in addition to parental consent)
* Patients not likely to survive the time period of the study washout period (4 months from enrolment)
* Treatment with an investigational drug or device within the last 3 months prior to enrolment
* Patients who are pregnant (a pregnancy test will be carried out for females of 11 years and above as is standard practice for clinical trials)
* Immediate families of investigators or site personnel directly affiliated with the study. Immediate family is defined as child or sibling, whether biological or legally adopted.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-05; Primary Completion 2012-12 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Biovolume of Pseudomonas Aeruginosa (PA) biofilms in sputum | 2 years
  Assessment of PA biofilms using FISH and image analysis, colony forming units and quantitative polymerase chain reaction.

SECONDARY OUTCOMES:
Bacterial density | 2 years
  To estimate the effect of adjunctive low dose inhaled nitric oxide given with standard antibiotic therapy on the whole community of bacteria within the CF lung by determination of CFU counts on non-selective agar.
Forced Expiratory Volume in 1 second (FEV1) | 2 years
  To assess the effect of NO on lung function measured by FEV1
Nitric Oxide levels in sputum | 2 years
  To estimate the NO levels in sputum in each group.
Bacterial species identification | 5 years
  To determine the characteristics in the wider microbial community within the CF lung using molecular methods during an exacerbation and to compare these characteristics between the two groups.
Exhaled Nitric Oxide | 2 years
  To assess the effect of low dose inhaled nitric oxide on exhaled nitric oxide levels
Health related quality of life score (HRQOL) | 2 years
  To assess the effect of low dose inhaled nitric oxide on HRQOL using the Cystic Fibrosis Questionnaire - United Kingdom (CFQ-UK).

CONTACTS AND LOCATIONS:
Overall Officials: Saul Faust, Principal Investigator — University Hopsital Southampton NHS Foundation Trust; Gary Connett, FRCPCH MD, Study Director — University Hospital Southampton NHS Foundation Trust; Jeremy Webb, PhD, Study Director — Universityh of Southampton
Locations (1):
- University Southampton NHS Foundation Trust, Southampton, Hampshire, United Kingdom

REFERENCES:
- See also: Published results — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5589160/